CLINICAL TRIAL: NCT02224261
Title: Effectiveness of Physical Therapy on Axillary Web Syndrome After Breast Cancer Surgery: a Randomized Controlled Trial
Brief Title: Effectiveness of Physical Therapy on Axillary Web Syndrome After Breast Cancer Surgery
Acronym: PTaws
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Collaborators: Hospital Universitario Principe de Asturias (Other)
Responsible Party: Principal Investigator, Maria Torres Lacomba, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11/032
Record Dates: First submitted 2014-08-20; First posted 2014-08-25 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Axillary Web Syndrome
Keywords: Axillary web syndrome; cording; physical therapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Therapy (Experimental): Physical therapy protocol includes manual lymph-drainage technique in axilla, and proximal ipsilateral arm, specific thumb manual lymph-drainage on the taut cords to make them gradually more flexible, in conjunction with progressive active and action-assisted arm exercises "stretching" cords and patient education.
  Interventions: Other: Physical Therapy protocol
- Control (Active Comparator): Control protocol includes standard progressive active and action-assisted arm exercises & patient education.
  Interventions: Other: Control

INTERVENTIONS:
Other: Physical Therapy protocol — Physical therapy protocol includes manual lymph-drainage technique in axilla, and proximal ipsilateral arm, specific thumb manual lymph-drainage on the taut cords to make them gradually more flexible, in conjunction with progressive active and action-assisted arm exercises "stretching" cords, and patient education.
  Other Names: PT-AWS
  Arms: Physical Therapy
Other: Control — Control protocol includes standard progressive active and action-assisted arm exercises & patient education.
  Other Names: CG
  Arms: Control

SUMMARY:
Objective: To determine the effectiveness of physical therapy on the axillary web syndrome in improving pain, reducing swelling and increasing mobility of the shoulder. Design: randomized single-blinded controlled trial. Follow-up: five physical therapy assessments: pre-intervention; post-intervention, 3 months post-intervention, 6 months post-intervention. Participants: Eighty consecutive women diagnosed with axillary web syndrome after undergoing unilateral breast cancer surgery with ALND or SLND at the Prıíncipe de Asturias Hospital in Alcalà de Henares, Madrid (Spain). Randomization: women will be randomly assigned to two groups by EpiData 3.1 software. Interventions: Physical Therapy group: Physical Therapy composed of manual lymph-drainage technique in axilla, and proximal ipsilateral arm, specific thumb manual lymph-drainage on the taut cords to make them gradually more flexible, in conjunction with progressive active and action-assisted arm exercises; Control group: standard progressive active and action-assisted arm exercises. 9 physical therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral breast cancer;
* Breast surgery with lymphadenectomy and / or sentinel lymph node biopsy;
* Axillary web syndrome in chest and / or upper limb of the operated side;
* VAS>3
* Consent to participate in the study;
* No contraindications for physical therapy (infection, metastasis);

Exclusion Criteria:

* Cognitive impairment;
* Visual impairment for reading;
* Lymphedema;
* Bilateral breast cancer;
* Systemic disease (metastases),
* Infection;
* Locoregional recurrence.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Subjective pain at one month (post-intervention); and 3 and 6 months post-intervention | Pre-intervention (baseline); Post-intervention (one month from baseline); and 3 and 6 months post-intervention
  Visual Analogue Scale

SECONDARY OUTCOMES:
Change from baseline in Range of shoulder motion at one month (post-intervention); and 3 and 6 months post-intervention | Pre-intervention (baseline); Post-intervention (one month from baseline); and 3 and 6 months post-intervention
  Inclinometer

OTHER OUTCOMES:
Change from baseline in QoL related to shoulder pain at one month (post-intervention); and 3 and 6 months post-intervention | Pre-intervention (baseline); Post-intervention (one month from baseline); and 3 and 6 months post-intervention
  Oxford Shoulder Score

CONTACTS AND LOCATIONS:
Locations (1):
- Physiotherapy in women´s health research group. University of Alcalà, Alcalà de Henares, Madrid, Spain

REFERENCES:
- [Background] Torres Lacomba M, Mayoral Del Moral O, Coperias Zazo JL, Yuste Sanchez MJ, Ferrandez JC, Zapico Goni A. Axillary web syndrome after axillary dissection in breast cancer: a prospective study. Breast Cancer Res Treat. 2009 Oct;117(3):625-30. doi: 10.1007/s10549-009-0371-8. Epub 2009 Mar 21. PMID 19306057
- [Result] Torres-Lacomba M, Prieto-Gomez V, Arranz-Martin B, Ferrandez JC, Yuste-Sanchez MJ, Navarro-Brazalez B, Romay-Barrero H. Manual Lymph Drainage With Progressive Arm Exercises for Axillary Web Syndrome After Breast Cancer Surgery: A Randomized Controlled Trial. Phys Ther. 2022 Mar 1;102(3):pzab314. doi: 10.1093/ptj/pzab314. PMID 35079831